CLINICAL TRIAL: NCT05765318
Title: Quadratus Lumborum Block for Total Abdominal Hysterectomy: a Double-blind, Randomized, Controlled Trial
Brief Title: Quadratus Lumborum Block for Total Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Center Niš (Other)
Responsible Party: Principal Investigator, Marija Kutlesic, MD Anaesthesiologoist, Principal investigator, Clinical Center Niš
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 150880200222
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Pain
Keywords: Quadratus lumborum block; Postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLB group (Experimental): At the end of surgery, before emergence of anesthesia, participants will receive bilateral QLB and intravenous (IV) ketoprofen 100 mg. Ketoprofen 100 mg IV will be repeated every 12 hours.
  For breakthrough pain patients will receive an IV bolus of morphine 5 mg. IV bolus can be repeated after 20 min. The maximum is 8 boluses for 4 hours.
  Interventions: Procedure: QLB
- Control group (No Intervention): At the end of surgery, before emergence of anesthesia, participants will receive IV ketoprofen 100 mg. Ketoprofen 100 mg IV will be repeated every 12 hours.
  For breakthrough pain patients will receive an IV bolus of morphine 5 mg. IV bolus can be repeated after 20 min. The maximum is 8 boluses for 4 hours.

INTERVENTIONS:
Procedure: QLB — QLB is ultrasound-guided injection of 30 ml bupivacaine 0.25% into quadratus lumborum plane posterior to the end of internal oblique muscle.
  Arms: QLB group

SUMMARY:
Procedure specific postoperative pain management (PROSPECT) guidelines for abdominal hysterectomy published in 2006 recommended laparoscopic or vaginal hysterectomy as a preferred surgical technique. Multimodal postoperative pain management plane includes cyclooxygenase-2 (COX-2) selective inhibitors, and/or conventional non-steroidal antiinflammatory drugs (NSAID) in combination with strong opioids for high-intensity pain or with weak opioids for moderate- or low-intensity pain. Paracetamol also was recommended in combination with COX-2 inhibitors or conventional NSAIDs. Epidural analgesia was recommended for high-risk patients. PROSPECT guidelines updated in 2018 discuss only perioperative approach for laparoscopic hysterectomy. However, hysterectomy technique has been switched from total abdominal to laparoscopic approach. In low resources settings, laparoscopic technique is nor well developed neither available to many patients. Furthermore, the majority of patients undergo total abdominal hysterectomy (TAH), that is very painful procedure. Quadratus lumborum block (QLB) is a regional analgesic technique described by Blanco in 2007. Society for Obstetric Anesthesiology and Perinatology (SOAP) and European Society for Regional Anaesthesia and Pain Therapy (ESRA) recommended QLB for post-Cesarean pain management in cases where intrathecal morphine could not be used or for breakthrough pain. Previous reports have shown that QLB is effective in providing pain relief after various abdominal operations. The effects of QLB for laparoscopic hysterectomy is controversial. We would like to see if QLB can provide analgesic benefits in multimodal pain management after TAH in our clinical settings.

DETAILED DESCRIPTION:
Participants will be randomly allocated into two groups. Experimental group will have QLB type 2 at the end of surgery, before emergence from general anesthesia. Control group will not have QLB.

All cases will be done under general anesthesia. During the surgery, the patients will be monitored with 5-lead electrocardiography, pulse oximetry, non-invasive blood pressure and end-expiratory CO2.

Standardized general anesthesia include induction with a propofol bolus of 1.5-2.5mg/kg and rocuronium 0.6mg/kg. Fentanyl 2 mcg/kg will be given at induction, and repeated to keep the blood pressure and heart rate changes up to 20% of baseline. Sevoflurane in a 50% air/50% oxygen mixture with an end-tidal of 1.5 vol% will be used as the maintenance agent. Mechanical ventilation will be maintained to keep the end-expiratory CO2 values between 34 and 36 mmHg. Incremental dose of rocuronium (0.15 mg/kg) will be given every 30 min or when needed. At the end of the surgery, after partial recovery from neuromuscular blockade, patients will receive atropine 0.01 mg/kg and neostigmine: 0.02mg/kg before tracheal extubation. Participants will be referred to the post-anesthesia recovery room after extubation and adequate hemodynamic and respiratory recovery.

Postoperative pain management will include ketoprofen and morphine.

ELIGIBILITY:
Inclusion Criteria:

1. endometrial carcinoma or uterine fibroids
2. American society of anesthesiologists (ASA) physical status 1-3,
3. Participant's body weight > 50 kg,
4. Written informed consent signed.

Exclusion Criteria:

1. Patient's refusal
2. Allergies to any study medication
3. Local skin infection on the site of QLB injection

3. Body mass index > 40 kg/m2 4. Inability to comprehend or participate in scoring scales 4. Deformations that could possibly affect the spread of the local anesthetic in the quadratus lumborum muscle plane 5. Quadratus lumborum muscle plane not seen in ultrasound examination 6. Patients on regular use of opioids 7. Psychiatric disorders

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants undergo total abdominal hysterectomy.
Enrollment: 60 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Morphine consumption (mg) during the first 12 postoperative hours | 12 hours after the end of surgery
  Total dose of IV morphine that participants received during the first 12 hours after surgery

SECONDARY OUTCOMES:
Pain at rest | 2, 6, 12, and 24 hours after surgery
  Pain at rest at NRS (Numeric rating scale score 0-10)
Pain at mobilization | 2, 6, 12, and 24 hours after surgery
  Pain at mobilization at NRS (Numeric rating scale score 0-10)
Cumulated morphine consumption (mg) at 24 hours postoperatively | 24 hours after the end of surgery
  Total dose of IV morphine that participants received during the first 24 hours after surgery
Time to first morphine demand | 24 hours after surgery
  Time to first request for rescue analgesia (morphine) after the end of surgery

OTHER OUTCOMES:
Postoperative nausea and vomiting (PONV) | 24 hours after surgery
  Recording PONV (Yes / No)

CONTACTS AND LOCATIONS:
Overall Officials: Nada Pejcic, M.D., Principal Investigator — Leskovac General Hospital
Locations (1):
- CCNis, Niš, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers engaging in independent scientific research could request data via email address: nada.pejcic@gmail.com
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact nada.pejcic@gmail.com

REFERENCES:
- [Background] Lirk P, Thiry J, Bonnet MP, Joshi GP, Bonnet F; PROSPECT Working Group. Pain management after laparoscopic hysterectomy: systematic review of literature and PROSPECT recommendations. Reg Anesth Pain Med. 2019 Apr;44(4):425-436. doi: 10.1136/rapm-2018-100024. Epub 2019 Feb 3. PMID 30914471
- [Background] Roofthooft E, Joshi GP, Rawal N, Van de Velde M; PROSPECT Working Group* of the European Society of Regional Anaesthesia and Pain Therapy and supported by the Obstetric Anaesthetists' Association. PROSPECT guideline for elective caesarean section: updated systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 May;76(5):665-680. doi: 10.1111/anae.15339. Epub 2020 Dec 28. PMID 33370462
- [Background] Bollag L, Lim G, Sultan P, Habib AS, Landau R, Zakowski M, Tiouririne M, Bhambhani S, Carvalho B. Society for Obstetric Anesthesia and Perinatology: Consensus Statement and Recommendations for Enhanced Recovery After Cesarean. Anesth Analg. 2021 May 1;132(5):1362-1377. doi: 10.1213/ANE.0000000000005257. PMID 33177330
- [Background] Akerman M, Pejcic N, Velickovic I. A Review of the Quadratus Lumborum Block and ERAS. Front Med (Lausanne). 2018 Feb 26;5:44. doi: 10.3389/fmed.2018.00044. eCollection 2018. PMID 29536008
- [Result] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Result] Hansen C, Dam M, Nielsen MV, Tanggaard KB, Poulsen TD, Bendtsen TF, Borglum J. Transmuscular quadratus lumborum block for total laparoscopic hysterectomy: a double-blind, randomized, placebo-controlled trial. Reg Anesth Pain Med. 2021 Jan;46(1):25-30. doi: 10.1136/rapm-2020-101931. Epub 2020 Oct 20. PMID 33082286
- [Derived] Pejcic N, Kutlesic M, Velickovic I, Milic V, Kovacevic S, Jankovic RJ, Mitic D, Mitic R, Zornic N. Quadratus lumborum block for total abdominal hysterectomy: a double-blind, randomized, controlled trial. Turk J Med Sci. 2025 Feb 7;55(2):349-359. doi: 10.55730/1300-0144.5978. eCollection 2025. PMID 40342315